CLINICAL TRIAL: NCT06039696
Title: Clinical Application of Pathogenic Metagenomic Next-generation Sequencing to Optimize the Diagnosis of Decompensated Cirrhosis Infection: a Multicenter, Prospective Study
Brief Title: Pathogenic Metagenomic Next-generation Sequencing to Optimize the Diagnosis of Decompensated Cirrhosis Infection
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-255
Record Dates: First submitted 2023-08-16; First posted 2023-09-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine, feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients received mNGS test: After enrolment, patients will receive mNGS test.

SUMMARY:
The goal of this observational study is to learn about clinical application of pathogenic metagenomic next-generation sequencing to optimize the diagnosis of infection in decompensated cirrhotic patients. The main questions it aims to answer are:

1. mNGS testing in optimizing anti-infective drug use in patients with acute decompensation, including response to empiric antibiotic therapy.
2. Proportion of patients with re-compensation.
3. The positive rate of mNGS in patients with acute decompensated cirrhosis and the characteristics of pathogen.
4. The incidence, risk factors and clinical correlation of CMV reactivation.

DETAILED DESCRIPTION:
Metagenomic next-generation sequencing (mNGS) is emerging as an important culture-independent technique that can detect nearly all known pathogens simultaneously from a clinical sample.Sequencing of microbial cell-free DNA (cfDNA) has recently been shown to enable diagnosis of several infection. Relevant studies on the clinical application of mNGS in cirrhosis patients are rare. The primary aim of this study was to comprehensively evaluate the fragments of genomic DNA from circulating microorganisms in acutely decompensated cirrhosis patients by sequencing the microbial cfDNA and relate this to clinical outcomes. The secondary aim was to validate the potential role of CMV reactivation, a known NHV with available antiviral medicines, in determining the prognosis of decompensated cirrhosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Diagnosis of cirrhosis, previously known or not, of any etiology, histologically proven or not.
* Acute decompensation: ascites, digestive hemorrhage or hepatic encephalopathy.

Exclusion Criteria:

* Age > 80 years old.
* Malignancy of liver or other organs (including leukemia).
* Receiving immunosuppressive agents for non-hepatic diseases.
* HIV infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diagnosis of cirrhosis hospitalized for acute decompensation
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Positive rate of mNGS test in AD patients | at enrolment

SECONDARY OUTCOMES:
90-day transplantation-free mortality | From enrollment to 90 days
Incidence of acute kidney injury (AKI) | From enrollment to 90 days
  AKI is defined as a change in SCr of ≥ 0.3 mg/dl (26.5 μmol/L) in ≤ 48 h, or a 50% increase in SCr from a baseline that is known or presumed to have occurred in the past 7 days.
Proportion of hospital readmissions due to infections | From enrollment to 90 days
Proportion of progression to SIRS or sepsis | From enrollment to 90 days
Consistency with blood culture results | at enrollment
  Concordance of mNGS With Other traditional Testing on Pathogens
Incidence of CMV reactivation | From enrollment to 90 days
  Cytomegalovirus DNA was quantified in stored plasma samples using real-time PCR (polymerase chain reaction) assay. DNA extraction was performed on 200 µL of plasma using a QIAamp DNA blood kit (Qiagen, German). Then, 25 µL of Tris (10 mM, pH 8.0) was used to elute the DNA, and 10 µL of the DNA was used for each PCR reaction. The minimum detection level was 102 copies/ml of plasma and values over this lower detection limit were considered to be CMV reactivation positive.
Rate of progression to acute-on-chronic liver failure (ACLF) | From enrollment to 90 days
  ACLF was defined according to the European Association for the Study of Liver-Chronic Liver Failure (EASL-CLIF) criteria. ACLF grade-1 includes three subgroups: 1) patients with single kidney failure; 2) patients with single failure of the liver, coagulation, circulation or respiration, who had serum creatinine ranging from 1.5 to 1.9 mg/dl and/or mild-to-moderate hepatic encephalopathy; and 3) patients with single cerebral failure who had serum creatinine ranging from 1.5 and 1.9 mg/dl. ACLF grade-2: patients with two organs failure. ACLF grade-3: patients with three organ failures or more. ACLF development: patients with absence of ACLF on admission and progression to ACLF within 28 days. The severity of liver disease was evaluated by the model of end-stage liver disease (MELD) score, Child-Pugh score and CLIF-AD score (in those without ACLF).

CONTACTS AND LOCATIONS:
Overall Officials: Chen Jinjun, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China